CLINICAL TRIAL: NCT01746251
Title: Randomized Phase II Study Comparing Concise Versus Prolonged Afatinib as Adjuvant Therapy for Patients With Resected Stage I-III NSCLC With EGFR Mutation
Brief Title: Adjuvant Afatinib in Stage I-III NSCLC With EGFR Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Lecia V. Sequist, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-504
Record Dates: First submitted 2012-11-27; First posted 2012-12-10 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: EGFR mutation; Resected
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concise Afatinib (Active Comparator): Afatinib oral daily dose for 3 months
  Interventions: Drug: Afatinib
- Prolonged Afatinib (Active Comparator): Afatinib oral daily dose for 2 years
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib

SUMMARY:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the drug is still being studied. It also means that the FDA has not yet approved afatinib for use in patients.

In this research study the investigators are looking to see if taking afatinib after surgery works better when taken over a short period of time, compared to a long period of time.

DETAILED DESCRIPTION:
In order to determine if one is eligible to participate in this study they would be asked to undergo some screening tests or procedures. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that one does not take part in the research study. If the patient has had some of these tests or procedures recently, they may or may not have to be repeated. These tests and procedures include: a medical history, performance status, physical exam and vital signs including height and weight, an assessment of your tumor, routine blood tests, pregnancy test, electrocardiogram, echocardiogram and/or multigated acquisition scan. If these tests show that a patient is eligible to participate in the research study, they will begin the study treatment. If one does not meet the eligibility criteria, they will not be able to participate in this research study.

Because no one knows which of the study options is best, the patients will be "randomized" into one of the study groups. They will take afatinib by mouth every day for either 3 months (short course) or for 2 years (long course). Randomization means that one is put into a group by chance. It is like flipping a coin. Neither the patient, nor the research doctor will choose what group the patient will be in. You will have a 50/50 chance of being placed in any group.

Regardless of which study group one is put in, all patients will take Afatinib by mouth every day. The first cycle will last 28 days. All cycles after that will last 25-31 days. Patients will take their medication (tablets) by mouth once a day, at about the same time each day. They should take Afatinib with a glass of water. Afatinib treatment will continue until the assigned course is completed, or until there are side effects that cannot be tolerated, or one decides to stop study treatment, of if the lung cancer returns.

Patients will be asked to come to the clinic at the following time points:

* Day 1 and 8 of Cycle 1
* Day 1 of Cycles 2, 3 and 4
* Off treatment visit-28 days after the last dose of study drug

If one is assigned to the long course, one will also need to come in for clinic visits on Day 1 of Cycles 7, 10, 13, 16, 19, 22 and 25. If one is assigned to the short course, one does not need to come in for these additional clinic visits.

The following tests and procedures will be done to monitor for side effects of afatinib.

* Routine blood tests-about 2 tablespoons of blood
* Performance status
* Physical exam and vital signs, including height and weight

The following tests and procedures will be done to monitor for recurrence of lung cancer. These visits are the same, regardless of whether one is taking a short course, or a long course of afatinib. There will be clinic visits once every 6 months for 3 years (months 7, 13, 19, 25, 31, 37 and 49), and then one more visit 1 year later. The following tests and procedures will be done at these follow up visits: a CT scan of the chest, routine blood tests, performance status and a physical exam, including height and weight.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of non-small cell lung cancer with EGFR mutation
* Complete surgical resection, pathologic stage IA-B, IIA-B, IIIA-B by AJCC 7th Edition staging criteria
* Surgical resection with curative intent was at least 6 months prior to enrollment
* At least 3 weeks have passed since completion of adjuvant chemotherapy or radiotherapy

Exclusion Criteria:

* Pregnant or breastfeeding
* History of allergic reactions attributed to compounds of similar chemical composition to afatinib
* Prior exposure to EGFR tyrosine kinase inhibitor
* Evidence of clinically active interstitial lung disease
* Radiographic evidence of recurrent NSCLC prior to afatinib treatment
* Receipt of any experimental treatment within 30 days of start of treatment with afatinib until the end of treatment visit
* Use of potent P-gp inhibitors and potent P-gp inducers must be avoided during treatment with afatinib
* Individuals with a history of a different malignancy (except: synchronous or metachronous primary non-small cell lung cancers of lower stage than the cancer for which adjuvant treatment is currently being prescribed; disease free for at least 3 years; cervical cancer in situ; basal or squamous cell carcinoma of the skin)
* HIV positive on combination antiretroviral therapy
* Uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2013-01; Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 2 years
  The primary objective of this study is to demonstrate that prolonged adjuvant therapy with afatinib will improve recurrence free survival (RFS) compared to a concise adjuvant course in patients with resected stage I-III non-small cell lung cancer (NSCLC) with epidermal growth factor receptor (EGFR) mutation.

SECONDARY OUTCOMES:
Number of patients with adverse events | 2 years
  To determine the safety and tolerability of adjuvant afatinib
Molecular genotype of recurrent cancers | 2 years
  We aim to collect clinical data from patients with recurrent NSCLC after treatment with adjuvant afatinib, including molecular characteristics of recurrent cancer analyzed as part of routine care, and time to treatment failure for patients treated with alternative chemotherapies for recurrent lung cancer.
overall survival | 2 years
  To estimate overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Lecia Sequist, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Stanford University, Palo Alto, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering, New York, New York